CLINICAL TRIAL: NCT00148577
Title: Pain Relief by Applying Transcutaneous Electrical Nerve Stimulation (TENS) on Acupuncture Points During the First Stage of Labour: a Randomised Controlled Trial
Brief Title: Pain Relief by Applying TENS on Acupuncture Points During the First Stage of Labour
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Other Study IDs: NMRPG1159
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Pain Relief at First Stage
Keywords: Pain Relief, TENS, Acupuncture Points
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
We aimed to establish the reduction of labor pain by applying TENS at acupuncture points during the first stage of labour, to assess their efficacy, and to ascertain their acceptability.

DETAILED DESCRIPTION:
We conducted a double-blind, placebo-controlled randomised trial involving healthy parturient at term pregnancy using TENS on 4 acupuncture points (Li 4 and Sp 6) (n=50) and the placebo group (n=50). Visual analogue scale (VAS) was used to assess the effect on pain before the application, 30 minutes and 60 minutes after TENS. The objective parameter of outcome was the score of VAS decreased in each groups. A post-partum questionnaire was given 24 hours later to evaluate the satisfaction and the use of this pain relieving method for the next delivery.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were:

* Voluntary informed participation to the study
* An initial wish to deliver without epidural analgesia
* Planned vaginal childbirth (non-obstetrical complicated pregnancy)
* Fetal vertex presentation
* Term pregnancy (>37 weeks of gestation)
* Apply at 1st stage of labour and excluded if cervical dilatation > 5 cm
* Age between 20 and 40 years
* Chinese speaking, capable to understand the study
* No experience of pain relief by systemic or epidural anesthesia in previous delivery
* No experience in acupuncture or TENS in other field
* Had no heart disease nor using pace-maker.

Exclusion Criteria:

* Cervical dilatation > 5 cm
* Experience of pain relief by systemic or epidural anesthesia in previous delivery
* Experience in acupuncture or TENS in other field
* Had heart disease or using pace-maker

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2002-08; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: An-Shine Chao, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan